CLINICAL TRIAL: NCT03308825
Title: Safety and Immunogenicity of Fluzone® Quadrivalent and Fluzone® High-Dose, Influenza Vaccines, 2017-2018 Formulations
Brief Title: Safety and Immunogenicity of Fluzone® Quadrivalent and Fluzone® High-Dose, Influenza Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC73; U1111-1183-5816 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2017-09-28; First posted 2017-10-13 (Actual); Results first posted 2018-12-17 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Influenza; Flu
Keywords: Influenza; Flu
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines

STUDY DESIGN:
Intervention Model Description: Multicenter, Open-label, Phase IV Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: 6 to < 36 Months (Experimental): Children aged 6 to < 36 months received a 0.25-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. For participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered on Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine
- Group 2: 3 to < 9 Years (Experimental): Children aged 3 to < 9 years received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0. For participants for whom 2 doses of influenza vaccine were recommended, a second dose was administered on Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine
- Group 3: 18 to < 65 Years (Experimental): Adults aged 18 to < 65 years received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone Quadrivalent vaccine
- Group 4: >= 65 Years (Experimental): Adults aged >= 65 years received a 0.5-mL dose of Fluzone High-Dose vaccine, intramuscularly, at Day 0.
  Interventions: Biological: Fluzone High-Dose vaccine

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine — 0.25 mL, Intramuscular
  Arms: Group 1: 6 to < 36 Months
Biological: Fluzone Quadrivalent vaccine — 0.5 mL, Intramuscular
  Arms: Group 2: 3 to < 9 Years; Group 3: 18 to < 65 Years
Biological: Fluzone High-Dose vaccine — 0.5 mL, Intramuscular
  Arms: Group 4: >= 65 Years

SUMMARY:
The aim of the study was to describe the safety and immunogenicity of the 2017-2018 formulation of Fluzone Quadrivalent vaccine in children 6 months to < 9 years of age, and in adults 18 to < 65 years of age, and to describe the safety and immunogenicity of the 2017-2018 formulation of Fluzone High-Dose vaccine in adults ≥ 65 years of age.

DETAILED DESCRIPTION:
All participants received 1 intramuscular dose of their assigned vaccine during Visit 1. For participants, for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP) guidance, a second dose of the same volume as the first dose was administered during Visit 2 (28 days after Visit 1). Solicited adverse reaction (AR) information was collected for 7 days following each vaccination. Unsolicited non-serious adverse event (AE) and serious adverse event (SAE) information was collected from Visit 1 to Visit 2 or from Visit 1 to Visit 3 for those participants receiving 2 doses of study vaccine.

Immunogenicity was evaluated in all participants prior to vaccination on Day 0 (Visit 1) and after the final vaccination (Day 28 post-final vaccination for participants 6 months to < 9 years of age and Day 21 post-vaccination for participants ≥ 18 years of age).

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months to < 9 years or ≥ 18 years on the day of first study vaccination (study product administration).
* For participants 6 to < 12 months of age, born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg (5.5 lbs).
* Informed consent form has been signed and dated by participants ≥ 18 years of age.
* Assent form was signed and dated by participants 7 to < 9 years of age, and informed consent form has been signed and dated by parent(s) or guardian(s) for participants 6 months to < 9 years of age.
* Participant and parent/guardian (of participants 6 months to < 9 years of age) were able to attend all scheduled visits and to comply with all study procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche, or post- menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure. Note: Participants may be considered eligible for enrollment if no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the participant would complete safety surveillance for the present study.
* Receipt of any vaccine in the 30 days preceding the first study vaccination, or planned receipt of any vaccine before Visit 2 for participants receiving 1 dose of influenza vaccine or Visit 3 for participants receiving 2 doses of influenza vaccine.
* Previous vaccination against influenza (in the 2017-2018 influenza season) with either study vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the 3 months preceding planned inclusion.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the 6 months preceding planned inclusion; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the 3 months preceding planned inclusion).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to study vaccine or to a vaccine containing any of the same substances. Note: The list of vaccine components is included in the Prescribing Information for each study vaccine.
* Thrombocytopenia, which may be a contraindication for intramuscular vaccination, at the discretion of the Investigator.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of planned vaccination or febrile illness (temperature ≥ 100.4 degree Fahrenheit [°F] [38.0 degrees Celsius {°C}]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study (participants ≥ 18 years of age) or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study (all participants).
* History of serious adverse reaction to any influenza vaccine.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- United States (3):
  - Sanofi Pasteur Investigational Site 003, Council Bluffs, Iowa
  - Sanofi Pasteur Investigational Site 002, Bardstown, Kentucky
  - Sanofi Pasteur Investigational Site 001, Metairie, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in 3 centers in the United States from 11 September 2017 to 25 October 2017.
Pre-assignment Details: A total of 240 participants were enrolled and vaccinated in the study.
Period: Overall Study
Arm/Group | Group 1: 6 to < 36 Months | Group 2: 3 to < 9 Years | Group 3: 18 to < 65 Years | Group 4: >= 65 Years
Started | 59 (1 child in Group 1 received a 0.5mL dose instead of a 0.25 mL dose and is included in Group 2.) | 61 (1 child in Group 1 received a 0.5mL dose instead of a 0.25 mL dose and is included in Group 2.) | 60 | 60
Completed | 57 | 57 | 59 | 60
Not Completed | 2 | 4 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis set included all participants who received at least 1 dose of study vaccine, according to the vaccine they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: 6 to < 36 Months | Group 2: 3 to < 9 Years | Group 3: 18 to < 65 Years | Group 4: >= 65 Years | Total
Number analyzed (Participants) | 59 | 61 | 60 | 60 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 61 | 1 | 0 | 121
  Between 18 and 65 years | 0 | 0 | 59 | 0 | 59
  >=65 years | 0 | 0 | 0 | 60 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 46 | 39 | 141
  Male | 34 | 30 | 14 | 21 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 0 | 1 | 10
  Not Hispanic or Latino | 56 | 55 | 60 | 59 | 230
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 29 | 30 | 16 | 5 | 80
  White | 29 | 25 | 43 | 53 | 150
  More than one race | 1 | 6 | 1 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site (Tenderness/Pain, Erythema, Swelling) and Systemic Reactions (Fever, Vomiting, Crying Abnormal, Drowsiness, Appetite Lost, Irritability): Group 1 (6 to < 36 Months)
Description: Solicited injection site reactions: Pain, Erythema and Swelling (Grade 3: Pain: cries when injected limb moved/ limb movement reduced, erythema and swelling >= 50 mm). Solicited systemic reactions: Fever, vomiting, abnormal crying, drowsiness, appetite lost, Irritability (Grade 3: Fever: >= 39.5 degrees Celsius [103.1 degree Fahrenheit {°F}], vomiting >= six episodes per 24 hours, abnormal crying : > 3 hours, drowsiness: sleeping most of the time or difficult to wake up, appetite lost: refuses >= 3 feeds/meals or refuses most feeds/meals, Irritability: Inconsolable).
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed using the Safety Analysis Set. Here, "Number analyzed" corresponds to participants with available data for each listed solicited reaction.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 6 to < 36 Months
Number analyzed (Participants) | 59
Participants
  Tenderness: number analyzed (Participants) | 56
  Tenderness | 16
  Tenderness : Grade 3: number analyzed (Participants) | 56
  Tenderness : Grade 3 | 1
  Erythema: number analyzed (Participants) | 56
  Erythema | 4
  Erythema : Grade 3: number analyzed (Participants) | 56
  Erythema : Grade 3 | 0
  Swelling: number analyzed (Participants) | 56
  Swelling | 2
  Swelling : Grade 3: number analyzed (Participants) | 56
  Swelling : Grade 3 | 0
  Fever: number analyzed (Participants) | 55
  Fever | 6
  Fever : Grade 3: number analyzed (Participants) | 55
  Fever : Grade 3 | 0
  Vomiting: number analyzed (Participants) | 56
  Vomiting | 2
  Vomiting : Grade 3: number analyzed (Participants) | 56
  Vomiting : Grade 3 | 0
  Crying Abnormal: number analyzed (Participants) | 56
  Crying Abnormal | 10
  Crying Abnormal : Grade 3: number analyzed (Participants) | 56
  Crying Abnormal : Grade 3 | 0
  Drowsiness: number analyzed (Participants) | 56
  Drowsiness | 11
  Drowsiness : Grade 3: number analyzed (Participants) | 56
  Drowsiness : Grade 3 | 0
  Appetite Lost: number analyzed (Participants) | 56
  Appetite Lost | 7
  Appetite Lost : Grade 3: number analyzed (Participants) | 56
  Appetite Lost : Grade 3 | 0
  Irritability: number analyzed (Participants) | 56
  Irritability | 13
  Irritability : Grade 3: number analyzed (Participants) | 56
  Irritability : Grade 3 | 0

2. Primary Outcome: Number of Participants Reporting Solicited Injection Site (Pain, Erythema, Swelling) and Systemic Reactions(Fever, Headache, Malaise, Myalgia): Group 2 (3 to < 9 Years), Group 3 (18 to < 65 Years) and Group 4(=< 65 Years)
Description: Solicited injection site reactions: Pain (Group 2: Grade 3: Incapacitating; Group 3 and 4: Grade 3: significant; prevents daily activity), erythema & swelling (Group 2: Grade 3: >= 50 mm, Group 3 and 4: Grade 3: > 100 mm). Solicited systemic reactions: Fever (Grade 3: >= 39.0 degrees Celsius [102.2°F]), headache, malaise & myalgia (Grade 3: significant interference with daily activities).
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed using Safety Analysis Set. Here, "Number analyzed" corresponds to participants with available data for each listed solicited reaction.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: 3 to < 9 Years | Group 3: 18 to < 65 Years | Group 4: >= 65 Years
Number analyzed (Participants) | 61 | 60 | 60
Participants
  Pain: number analyzed (Participants) | 56 | 58 | 60
  Pain | 25 | 27 | 20
  Pain: Grade 3: number analyzed (Participants) | 56 | 58 | 60
  Pain: Grade 3 | 1 | 1 | 0
  Erythema: number analyzed (Participants) | 57 | 58 | 60
  Erythema | 9 | 0 | 3
  Erythema : Grade 3: number analyzed (Participants) | 57 | 58 | 60
  Erythema : Grade 3 | 3 | 0 | 0
  Swelling: number analyzed (Participants) | 57 | 58 | 60
  Swelling | 11 | 1 | 2
  Swelling : Grade 3: number analyzed (Participants) | 57 | 58 | 60
  Swelling : Grade 3 | 2 | 0 | 0
  Fever: number analyzed (Participants) | 56 | 58 | 60
  Fever | 1 | 0 | 1
  Fever : Grade 3: number analyzed (Participants) | 56 | 58 | 60
  Fever : Grade 3 | 1 | 0 | 1
  Headache: number analyzed (Participants) | 56 | 58 | 60
  Headache | 2 | 10 | 6
  Headache : Grade 3: number analyzed (Participants) | 56 | 58 | 60
  Headache : Grade 3 | 0 | 1 | 0
  Malaise: number analyzed (Participants) | 56 | 58 | 60
  Malaise | 3 | 5 | 9
  Malaise: Grade 3: number analyzed (Participants) | 56 | 58 | 60
  Malaise: Grade 3 | 1 | 1 | 0
  Myalgia: number analyzed (Participants) | 56 | 58 | 60
  Myalgia | 11 | 13 | 17
  Myalgia : Grade 3: number analyzed (Participants) | 56 | 58 | 60
  Myalgia : Grade 3 | 0 | 1 | 1

3. Primary Outcome: Geometric Mean Titers (GMTs) of Influenza Vaccine Antibodies in Children: Group 1 (6 to < 36 Months) and Group 2 (3 to < 9 Years)
Description: Anti-influenza antibodies were measured using the hemagglutination inhibition (HAI) assay for 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Per-Protocol Analysis Set (PPAS) included all participants who received at least 1dose of study vaccine, had a valid post-final vaccination serology result for at least 1 strain and did not have any major protocol deviations. Here, "Number analyzed" corresponds to participants with available data for each listed strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Group 1: 6 to < 36 Months | Group 2: 3 to < 9 Years
Number analyzed (Participants) | 52 | 55
Titers (1/dilutions)
  Pre-Vaccination: A/H1N1: number analyzed (Participants) | 51 | 55
  Pre-Vaccination: A/H1N1 | 19.9 [11.9 to 33.1] | 306 [198 to 473]
  Pre-Vaccination: A/H3N2: number analyzed (Participants) | 51 | 52
  Pre-Vaccination: A/H3N2 | 49.7 [27.7 to 89.2] | 415 [253 to 681]
  Pre-Vaccination: B Victoria: number analyzed (Participants) | 50 | 55
  Pre-Vaccination: B Victoria | 32.0 [19.7 to 52.0] | 180 [112 to 290]
  Pre-Vaccination: B Yamagata: number analyzed (Participants) | 50 | 55
  Pre-Vaccination: B Yamagata | 43.5 [27.6 to 68.5] | 334 [219 to 510]
  Post-Final Vaccination: A/H1N1 | 450 [301 to 671] | 1606 [1198 to 2153]
  Post-Final Vaccination: A/H3N2: number analyzed (Participants) | 52 | 54
  Post-Final Vaccination: A/H3N2 | 568 [336 to 958] | 2370 [1712 to 3282]
  Post-Final Vaccination: B Victoria | 481 [313 to 738] | 1668 [1142 to 2436]
  Post-Final Vaccination: B Yamagata | 698 [465 to 1047] | 2187 [1610 to 2971]

4. Primary Outcome: GMTs of Influenza Vaccine Antibodies in Adults: Group 3 (18 to < 65 Years) and Group 4 (>= 65 Years)
Description: Anti-influenza antibodies were measured using the HAI assay for each of the following 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage (for Group 3) and for 3 strains: H1N1, H3N2, and B Victoria lineage (for Group 4).
Time Frame: Day 0 (pre-vaccination) and Day 21 (post-vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed" corresponds to participants with available data for each listed strain and "0" in the number analyzed field signifies that none of the participants were analyzed, since the 2017-2018 formulation of Fluzone High-Dose vaccine did not contain the B Yagamata lineage strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilutions)
Arm/Group | Group 3: 18 to < 65 Years | Group 4: >= 65 Years
Number analyzed (Participants) | 56 | 59
Titers (1/dilutions)
  Pre-Vaccination: A/H1N1: number analyzed (Participants) | 55 | 59
  Pre-Vaccination: A/H1N1 | 165 [110 to 248] | 74.6 [52.3 to 106]
  Pre-Vaccination: A/H3N2: number analyzed (Participants) | 53 | 59
  Pre-Vaccination: A/H3N2 | 231 [150 to 356] | 194 [130 to 291]
  Pre-Vaccination: B Victoria | 276 [185 to 412] | 215 [151 to 305]
  Pre-Vaccination: B Yamagata: number analyzed (Participants) | 55 | 0
  Pre-Vaccination: B Yamagata | 425 [308 to 587] |
  Post-Final Vaccination: A/H1N1 | 756 [539 to 1062] | 393 [275 to 561]
  Post-Final Vaccination: A/H3N2: number analyzed (Participants) | 55 | 59
  Post-Final Vaccination: A/H3N2 | 1128 [791 to 1610] | 864 [612 to 1218]
  Post-Final Vaccination: B Victoria | 1117 [853 to 1463] | 644 [465 to 892]
  Post-Final Vaccination: B Yamagata: number analyzed (Participants) | 56 | 0
  Post-Final Vaccination: B Yamagata | 1312 [1010 to 1704] |

5. Primary Outcome: GMT Ratios (GMTRs) of Influenza Vaccine Antibodies in Children: Group 1 (6 to < 36 Months) and Group 2 (3 to < 9 Years)
Description: GMTRs are the geometric means of the individual post-final vaccination/pre-vaccination titer ratios for each of the following 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage, measured using the HAI assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-final vaccination)
Population: Analysis was performed on PPAS. Here, "Number analyzed" corresponds to participants with available data for each listed strain.
Measure: Number (95% Confidence Interval); unit: Titer Ratio
Arm/Group | Group 1: 6 to < 36 Months | Group 2: 3 to < 9 Years
Number analyzed (Participants) | 52 | 55
Titer Ratio
  A/H1N1: number analyzed (Participants) | 51 | 55
  A/H1N1 | 17.6 [12.1 to 25.6] | 5.05 [3.56 to 7.16]
  A/H3N2: number analyzed (Participants) | 51 | 52
  A/H3N2 | 10.8 [7.54 to 15.4] | 5.54 [3.67 to 8.37]
  B Victoria: number analyzed (Participants) | 50 | 55
  B Victoria | 13.1 [8.86 to 19.3] | 9.02 [6.06 to 13.4]
  B Yamagata: number analyzed (Participants) | 50 | 55
  B Yamagata | 14.0 [9.44 to 20.8] | 6.46 [4.70 to 8.88]

6. Primary Outcome: GMTRs of Influenza Vaccine Antibodies in Adults: Group 3 (18 to < 65 Years) and Group 4 (>= 65 Years)
Description: GMTRs are the geometric means of the individual post-final vaccination/pre-vaccination titer ratios for each of the following 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage (for Group 3) and for 3 strains: H1N1, H3N2, and B Victoria lineage (for Group 4), measured using the HAI assay.
Time Frame: Day 0 (pre-vaccination) and Day 21 (post-vaccination)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Titer Ratio
Groups:
- Group 4: Adults >= 65 Years: Adults >= 65 years of age received an intramuscular 0.5-mL dose of Fluzone High-Dose vaccine on Day 0.
Arm/Group | Group 3: 18 to < 65 Years | Group 4: Adults >= 65 Years
Number analyzed (Participants) | 56 | 59
Titer Ratio
  A/H1N1: number analyzed (Participants) | 55 | 59
  A/H1N1 | 4.31 [2.91 to 6.40] | 5.15 [3.50 to 7.57]
  A/H3N2: number analyzed (Participants) | 53 | 59
  A/H3N2 | 4.44 [2.88 to 6.85] | 4.45 [3.09 to 6.40]
  B Victoria | 4.05 [2.55 to 6.43] | 2.96 [2.26 to 3.88]
  B Yamagata: number analyzed (Participants) | 55 | 0
  B Yamagata | 3.09 [2.16 to 4.42] |

7. Primary Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens: Group 1 (6 to < 36 Months) and Group 2 (3 to < 9 Years)
Description: Anti-influenza antibodies were measured using the HAI assay for 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage. Seroprotection was defined as antibody titer >=40 (1/ dilution) at pre-vaccination or at post-final vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 6 to < 36 Months | Group 2: 3 to < 9 Years
Number analyzed (Participants) | 52 | 55
Participants
  Pre-Vaccination: A/H1N1: number analyzed (Participants) | 51 | 55
  Pre-Vaccination: A/H1N1 | 15 | 48
  Pre-Vaccination: A/H3N2: number analyzed (Participants) | 51 | 52
  Pre-Vaccination: A/H3N2 | 24 | 46
  Pre-Vaccination: B Victoria: number analyzed (Participants) | 50 | 55
  Pre-Vaccination: B Victoria | 21 | 44
  Pre-Vaccination: B Yamagata: number analyzed (Participants) | 50 | 55
  Pre-Vaccination: B Yamagata | 31 | 50
  Post-Final Vaccination: A/H1N1 | 51 | 54
  Post-Final Vaccination: A/H3N2: number analyzed (Participants) | 52 | 54
  Post-Final Vaccination: A/H3N2 | 50 | 54
  Post-Final Vaccination: B Victoria | 50 | 54
  Post-Final Vaccination: B Yamagata | 50 | 55

8. Primary Outcome: Number of Participants With Seroprotection to Influenza Vaccine Antigens: Group 3 (18 to < 65 Years) and Group 4 (>= 65 Years)
Description: Anti-influenza antibodies were measured using the HAI assay for each of the following 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage (for Group 3) and for 3 strains: H1N1, H3N2, and B Victoria lineage (for Group 4). Seroprotection was defined as antibody titer >= 40 (1/ dilution) at pre-vaccination or at post-final vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 21 (post-vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: 18 to < 65 Years | Group 4: >= 65 Years
Number analyzed (Participants) | 56 | 59
Participants
  Pre-Vaccination: A/H1N1: number analyzed (Participants) | 55 | 59
  Pre-Vaccination: A/H1N1 | 45 | 40
  Pre-Vaccination: A/H3N2: number analyzed (Participants) | 53 | 59
  Pre-Vaccination: A/H3N2 | 48 | 49
  Pre-Vaccination: B Victoria | 48 | 55
  Pre-Vaccination: B Yamagata: number analyzed (Participants) | 55 | 0
  Pre-Vaccination: B Yamagata | 54 |
  Post-Final Vaccination: A/H1N1 | 55 | 57
  Post-Final Vaccination: A/H3N2: number analyzed (Participants) | 55 | 59
  Post-Final Vaccination: A/H3N2 | 55 | 59
  Post-Final Vaccination: B Victoria | 56 | 58
  Post-Final Vaccination: B Yamagata: number analyzed (Participants) | 56 | 0
  Post-Final Vaccination: B Yamagata | 56 |

9. Primary Outcome: Number of Participants With Seroconversion to Influenza Vaccine Antigens: Group 1 (6 to < 36 Months) and Group 2 (3 to < 9 Years)
Description: Anti-influenza antibodies were measured using the HAI assay for 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage. Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-final vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and at least a 4-fold increase in post-final vaccination titer.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-final vaccination)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: 6 to < 36 Months | Group 2: 3 to < 9 Years
Number analyzed (Participants) | 52 | 55
Participants
  A/H1N1: number analyzed (Participants) | 51 | 55
  A/H1N1 | 45 | 28
  A/H3N2: number analyzed (Participants) | 51 | 52
  A/H3N2 | 42 | 30
  B Victoria: number analyzed (Participants) | 50 | 55
  B Victoria | 44 | 39
  B Yamagata: number analyzed (Participants) | 50 | 55
  B Yamagata | 46 | 36

10. Primary Outcome: Number of Participants With Seroconversion to Influenza Vaccine Antigens: Group 3 (18 to < 65 Years) and Group 4 (>= 65 Years)
Description: Anti-influenza antibodies were measured using the HAI assay for each of the following 4 strains: H1N1, H3N2, B Victoria lineage, and B Yamagata lineage (for Group 3) and for 3 strains: H1N1, H3N2, and B Victoria lineage (for Group 4). Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-final vaccination titer >= 1:40 or a pre-vaccination titer >= 1:10 and at least a 4-fold increase in post-final vaccination titer.
Time Frame: Day 0 (pre-vaccination) and Day 21 (post-vaccination)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: 18 to < 65 Years | Group 4: >= 65 Years
Number analyzed (Participants) | 56 | 59
Participants
  A/H1N1: number analyzed (Participants) | 55 | 59
  A/H1N1 | 26 | 33
  A/H3N2: number analyzed (Participants) | 53 | 59
  A/H3N2 | 22 | 33
  B Victoria | 19 | 18
  B Yamagata: number analyzed (Participants) | 55 | 0
  B Yamagata | 22 |

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to Day 56 for Groups 1 and 2; up to Day 21 for Groups 3 and 4.
Description: A solicited reaction is an AE that is prelisted in the electronic case report form (eCRF) and considered to be related to vaccination. A solicited reaction is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature and time to onset) prelisted (i.e., solicited) in the eCRF. An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or time to onset post-vaccination.
Arm/Group | Group 1: 6 to < 36 Months | Group 2: 3 to < 9 Years | Group 3: 18 to < 65 Years | Group 4: >= 65 Years
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/61 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61 | 2/60 | 0/60
Other Adverse Events (participants affected / at risk) | 30/59 | 30/61 | 29/60 | 30/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 6 to < 36 Months (N=59) | Group 2: 3 to < 9 Years (N=61) | Group 3: 18 to < 65 Years (N=60) | Group 4: >= 65 Years (N=60)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: 6 to < 36 Months (N=59) | Group 2: 3 to < 9 Years (N=61) | Group 3: 18 to < 65 Years (N=60) | Group 4: >= 65 Years (N=60)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Crying (General disorders) | 10 (11) | 1 (1) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 4 (4) | 9 (9) | 0 (0) | 3 (3)
Injection Site Pain (General disorders) | 16 (18) | 26 (26) | 27 (27) | 20 (20)
Injection Site Swelling (General disorders) | 2 (2) | 11 (11) | 1 (1) | 2 (2)
Malaise (General disorders) | 0 (0) | 3 (3) | 5 (5) | 9 (9)
Pyrexia (General disorders) | 8 (9) | 2 (2) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (11) | 13 (13) | 17 (17)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 10 (10) | 7 (7)
Somnolence (Nervous system disorders) | 11 (13) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 13 (13) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT03308825/Prot_001.pdf
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03308825/SAP_000.pdf